CLINICAL TRIAL: NCT02720341
Title: Virtual, Intensified and Patient-tailored Robotic Arm Therapy With the Exoskeleton Robot ARMin
Brief Title: VIT-ARMin Virtual, Intensified and Patient-tailored Robotic Arm Therapy With the Exoskeleton Robot ARMin
Acronym: VIT-ARMin
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Doctoral students on project defended their thesis.
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Klinik Lengg, Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VIT-ARMin
Record Dates: First submitted 2016-02-11; First posted 2016-03-25 (Estimated); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Stroke; Spinal Cord Injury; Healthy
MeSH Terms: conditions — Stroke; Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ARMin (Experimental): Therapy on ARMin robotic device
  Interventions: Device: ARMin

INTERVENTIONS:
Device: ARMin — single sessions of about one hour each

SUMMARY:
Consideration-of-Concept Trial (stage 1) on robotic therapy of the upper extremity with the ARMin therapy robot in healthy subjects and patients with neurological disease (e.g. stroke, spinal cord injury)

DETAILED DESCRIPTION:
Neurological patients (e.g., after stroke) need long-term neurorehabilitative therapy of the arm with often limited, unsatisfactory outcome. Robots became a promising supplement or even alternative for neurorehabilitative training. Investigators aim at developing a unique intensified and patient-tailored robot-aided training strategy of the arm. The exoskeleton robot ARMin will be further developed to adapt software components accordingly. The goal is to enhance treatment efficacy to an extent that the improvement in motor function is meaningful for the individual patient. It can be intensified by different strategies that will be evaluated alone and in combination. These strategies include:

strength training an error-amplification strategy increased number of repetitions multisensory feedback multiplayer approach

ELIGIBILITY:
Inclusion Criteria:

healthy or CVA or spinal cord injury

* Aged ≥18 years
* No excessive spasticity of the affected arm (modified Ashworth Scale ≤3)
* No serious medical or psychiatric disorder as assessed by their physician
* No orthopaedic, rheumatological, or other disease restricting movements of the paretic arm
* No shoulder subluxation (palpation <2 fingers)
* No skin ulcerations at the paretic arm
* Ability to communicate effectively with the examiner such that the validity of the patient's data could not be compromised
* No cybersickness (e.g., nausea when looking at a screen or playing computer games)
* No pacemaker or other implanted electric devices
* Bodyweight <120 kg
* No serious cognitive defects or aphasia preventing effective use of ARMin

Exclusion Criteria

- Allergy against alcohol or no agreement for skin shaving

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2015-04-10 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Intrinsic Motivation Inventory (IMI) questionaire | within one day
  The IMI is a multidimensional measurement device that assesses participants' interest/enjoyment, perceived competence, effort, value/usefulness, felt pressure and tension, and perceived choice while performing a given activity, thus yielding six subscale scores

SECONDARY OUTCOMES:
performance tests (kinematic and kinetic data) in virtual reality on the ARMin robot (time in msec) | within one day
  kinematic and kinetic data during motor performance will be recorded
performance tests (kinematic and kinetic data) in virtual reality on the ARMin robot (position in cm) | within one day
  kinematic and kinetic data during motor performance will be recorded
performance tests (kinematic and kinetic data) in virtual reality on the ARMin robot ( force in Nm) | within one day
  kinematic and kinetic data during motor performance will be recorded
muscle strength in Nm | within one day
  muscle strength will be recorded by the device
questionaire on interaction, time and effort | within one day
  questions rated on a analog scale by the participant regarding the interaction with participants and therapists, the perceived time and the perceived effort
EMG for muscle activity (time and electric potential) | within one day
  The level of muscular activity will be assessed by surface electromyography (EMG). The EMG device to be employed is a wireless commercially available certified device (Noraxon). EMG activity of different shoulder and elbow muscles will be recorded using surface electrodes to compare muscle activations in different muscles
EMG for muscle activity (time in sec) | within one day
  The level of muscular activity will be assessed by surface electromyography (EMG). The EMG device to be employed is a wireless commercially available certified device (Noraxon). EMG activity of different shoulder and elbow muscles will be recorded using surface electrodes to compare muscle activations in different muscles
EMG for muscle activity (electric potential in V) | within one day
  The level of muscular activity will be assessed by surface electromyography (EMG). The EMG device to be employed is a wireless commercially available certified device (Noraxon). EMG activity of different shoulder and elbow muscles will be recorded using surface electrodes to compare muscle activations in different muscles
detection thresholds (time) | within one day
  Detection thresholds for sensory stimuli will be assessed
detection thresholds (position in cm) | within one day
  Detection thresholds for sensory stimuli will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Robert Riener, PhD, Study Chair — ETH Zurich
Locations (3):
- Switzerland (3):
  - Labor für Sensomotorische Systeme, ETH Zürich, Balgrist Campus, Zurich
  - Balgrist Campus, Zurich
  - Klinik Lengg, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aghamohammadi NR, Bittmann MF, Klamroth-Marganska V, Riener R, Huang FC, Patton JL. Error fields: personalized robotic movement training that augments one's more likely mistakes. Sci Rep. 2025 Feb 4;15(1):4201. doi: 10.1038/s41598-025-87331-x. PMID 39905053
- [Derived] Just F, Ozen O, Tortora S, Klamroth-Marganska V, Riener R, Rauter G. Human arm weight compensation in rehabilitation robotics: efficacy of three distinct methods. J Neuroeng Rehabil. 2020 Feb 5;17(1):13. doi: 10.1186/s12984-020-0644-3. PMID 32024528
- [Derived] Baur K, Speth F, Nagle A, Riener R, Klamroth-Marganska V. Music meets robotics: a prospective randomized study on motivation during robot aided therapy. J Neuroeng Rehabil. 2018 Aug 16;15(1):79. doi: 10.1186/s12984-018-0413-8. PMID 30115082